CLINICAL TRIAL: NCT02962206
Title: The Effect of Point-of-care Ultrasound Guidance for Distal Radius Fracture Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcus Van Aarsen (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor-Investigator, Marcus Van Aarsen, Resident Physician, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107331
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Point-of-care Ultrasound, Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Closed Fracture Reduction

ARMS (2):
- Standard of care (Active Comparator): Patients will undergo standard closed fracture reduction. The sedation type, reduction method, and immobilization method will be at the discretion of the treating physician. Point-of-care ultrasound will not be used.
  Interventions: Procedure: Closed fracture reduction
- Experimental Group (Experimental): Patients will undergo standard closed fracture reduction with the addition of point-of-care ultrasound use to assess post-reduction dorsal angulation. The sedation type, reduction method, and immobilization method will be at the discretion of the treating physician.
  Interventions: Device: Point-of-care ultrasound; Procedure: Closed fracture reduction

INTERVENTIONS:
Device: Point-of-care ultrasound — After the fracture reduction maneouver, the physician will assess residual dorsal angulation using point-of-care ultrasound. If deemed adequate, the physician will progress to immobilization. If the reduction is not adequate, the physician will attempt further reduction at their discretion.
  Other Names: POCUS
  Arms: Experimental Group
Procedure: Closed fracture reduction — The distal radius fracture will be reduced with using a combination of local anesthetic, sedation, reduction maneouvers and immobiliazation at the discretion of the treating physician

SUMMARY:
Distal radius (Colle's) fractures in adult patients are commonly reduced in the emergency department before casting. Standard of care currently requires that x-rays be performed before and after fracture reduction, and inadequate reductions may be subject to repeat attempts and are at a higher risk to require surgery. This study will assess the use of point-of-care ultrasound (POCUS) in addition to standard care as a tool to decrease the angulation at the fracture site after a reduction is performed. If this angulation is decreased, it would suggest that POCUS for distal radius fracture reduction could decrease the number of failed reduction attempts and therefore the number of repeated reduction attempts.

ELIGIBILITY:
Inclusion Criteria:

* radiographically confirmed distal radius fracture

Exclusion Criteria:

* patients who do not consent
* patients with multiple acute injuries, open fractures, or other local fractures evident (a simple ulnar styloid fracture will not be considered an exclusion criterion)
* patients with neurovascular compromise
* patients with bilateral distal radius fractures
* patients with minimally displaced distal radius fractures that do not require closed reduction before casting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Residual dorsal angulation | Collected at the same-day post-reduction xray. Data will be aggregated over 1 year

SECONDARY OUTCOMES:
Need for orthopaedic surgery within 6 weeks of injury | To be assessed 6 weeks post-injury. Data will be aggregated over the 1 year study period
  To be acquired via electronic patient charting
Physician satisfaction: post-reduction questionnaire | Questionnaire to be administered immediately after reduction. Data to be aggregated during the 1 year study period

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Health Care London, London, Ontario
  - London Health Sciences Centre, London, Ontario